CLINICAL TRIAL: NCT00684970
Title: A Phase IIB Clinical Trial of the Anti-Angiogenic Drug Combination Hamsa-1™ in Metastatic Castration Resistant Prostate Cancer (CRPC)
Brief Title: Phase IIB Clinical Trial of Hamsa-1™ in Metastatic Castration Resistant Prostate Cancer (CRPC)
Acronym: TLH-202
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tiltan Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLH-202
Record Dates: First submitted 2008-05-22; First posted 2008-05-28 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Metastatic Castration Resistant Prostate Cancer (CRPC)
Keywords: CRPC; HRPC; metastatic prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hamsa-1™ TL-118 (Other): Once daily Hamsa-1™ TL-118 (single arm)
  Interventions: Drug: Hamsa-1™ TL-118

INTERVENTIONS:
Drug: Hamsa-1™ TL-118 — Once daily Hamsa-1™ TL-118

SUMMARY:
Hamsa-1™ is an anti-angiogenic drug combination designed for the treatment of cancer. The investigational product Hamsa-1™ comprises of four well-known active components. The therapy is administrated at a unique dosing regimen that was found to be effective and advantageous in terms of safety.The product is formulated as an oral suspension, conveniently administrated by the patients at home and not requiring medical staff assistance. This Phase IIb clinical trial aims to evaluate the efficacy of Hamsa-1™ for the treatment of metastatic Castration Resistant Prostate Cancer (CRPC) patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects willing and able to give written informed consent
2. Confirmed metastatic castration resistant prostate cancer and rising PSA
3. ECOG performance status ≤ 1
4. Adequate renal function, hepatic function and bone marrow reserve.
5. Subjects capable of swallowing.

Exclusion Criteria:

1. Hypersensitivity to one or more of the Hamsa-1™ active components
2. Glucose-6-phosphate-dehydrogenase deficiency (G6PD)
3. Subjects with a clinically significant or unstable medical condition that would preclude safe and complete study participation
4. Subjects who received any investigational medication, antineoplastic therapy, or any significant change in treatment within 1 month prior to screening
5. Subjects with visceral metastases (e.g. liver, lung)
6. Subjects who received more than 2 prior chemotherapies for the treatment of prostate cancer
7. Subjects suffering from circumstances likely to interfere with absorption of orally administrated drugs
8. Subjects unwilling to or unable to comply with study protocol

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-03; Primary Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) measured 24 weeks after treatment initiation | 24 weeks and up to 3 years

SECONDARY OUTCOMES:
Overall Survival, Time to PSA Progression, PSA Response, Pain Response measured in evaluable patients. | 52 weeks and up to 3 years
Safety and tolerability | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Dan Goldstaub, PhD, Study Director — Chief Operating Officer, Tiltan Pharma LtD
Locations (5):
- Israel (5):
  - Bnei Tzion Medical Center, Haifa
  - Rambam Medical Center, Haifa
  - Sourasky Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky
  - Asaf Harofe Medical Center, Tzrifin